CLINICAL TRIAL: NCT01548339
Title: Laparoscopic Cholecystectomy for Acute Cholecystitis: is the Rule of 72 Hours Still Actual?
Brief Title: Laparoscopic Cholecystectomy for Acute Cholecystitis After 72 Hours of Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermediary analysis showing increased morbidity in the delayed group
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Chairman of the Department of Surgery, Professor of Surgery, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 252/08 CHV
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Acute Cholecystitis; Cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed (Active Comparator): Laparoscopic cholecystectomy performed secondarily after an initial conservative treatment
  Interventions: Procedure: Laparoscopic cholecystectomy
- Early (Experimental): Laparoscopic cholecystectomy performed directly after the initial diagnosis
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — 3 trocars laparoscopic cholecystectomy

SUMMARY:
The purpose of this study is to compare the clinical outcomes of early versus delayed laparoscopic cholecystectomies for acute cholecystitis with more than 72 hours of symptoms.

DETAILED DESCRIPTION:
In acute biliary cholecystitis, there was a dogma that patients should be operated within 72 hours of evolution. However, retrospective studies suggested that laparoscopic cholecystectomy even after 72 hours was safe. Moreover, some randomized controlled-trials did not found any differences in term of complications between early and delayed cholecystectomy, however none of these studies did separate patients according to the onset of symptoms. The aim of our present study was to compare the clinical outcomes of immediate versus delayed cholecystectomies for acute cholecystitis with more than 72 hours of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* proven echographic cholecystitis

Exclusion Criteria:

* pregnancy
* immunosuppression
* severe sepsis
* perforated cholecystitis
* peritonitis
* cholangitis
* acute pancreatitis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-02; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Demartines, MD, Study Chair — University of Lausanne Hospitals; Nermin Halkic, MD, Study Director — University of Lausanne Hospitals; Luca Di Mare, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Roulin D, Saadi A, Di Mare L, Demartines N, Halkic N. Early Versus Delayed Cholecystectomy for Acute Cholecystitis, Are the 72 hours Still the Rule?: A Randomized Trial. Ann Surg. 2016 Nov;264(5):717-722. doi: 10.1097/SLA.0000000000001886. PMID 27741006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed | Early
Started | 44 | 42
Completed | 38 | 41
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed | Early | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (16.6) | 55.8 (16.8) | 56.9 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  Switzerland | 44 | 42 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event ("Global Morbidity").
Description: any adverse event occurring from time of diagnosis until the 30th postoperative day
Time Frame: 30 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed | Early
Number analyzed (Participants) | 44 | 42
Participants | 17 | 6

2. Secondary Outcome: Postoperative Complications
Description: postoperative complications graded according to Clavien classification
Time Frame: 30 postoperative days
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed | Early
Number analyzed (Participants) | 44 | 42
Participants | 7 | 6

3. Secondary Outcome: Length of Stay
Description: total in hospital stay
Time Frame: 30 postoperative days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Delayed | Early
Number analyzed (Participants) | 44 | 42
days | 7 [5 to 11] | 4 [3 to 4]

ADVERSE EVENTS:
Arm/Group | Delayed | Early
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/44 | 2/42
Other Adverse Events (participants affected / at risk) | 4/44 | 4/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed (N=44) | Early (N=42)
postoperative choledocolithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
pulmonary acute oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
biliary leak (Hepatobiliary disorders) | 1 (1) | 0 (0)
anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed (N=44) | Early (N=42)
surgical site infection (Surgical and medical procedures) | 3 (3) | 3 (3)
urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes